CLINICAL TRIAL: NCT00698997
Title: Intensive Intervention for Toddlers With Autism
Brief Title: Intensive Intervention for Toddlers With Autism (EARLY STEPS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of Washington (Other); University of Michigan (Other); National Institutes of Health (NIH) (NIH); University of California, Los Angeles (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200816233; 1R01MH081757 (NIH)
Record Dates: First submitted 2008-06-12; First posted 2008-06-17 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: autism; autism spectrum disorder; intensive intervention for toddlers with autism; PDD NOS; early steps study; early start denver model; early intervention for infants and toddlers with autism; toddler treatment; Sally Rogers; University of California, Davis; University of Michigan; MIND Institute
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Early Start Denver Model (Experimental): Phase 1 of ESDM intervention: 12 weekly, 1 to 1.5 hr. sessions focused on teaching & coaching parents to use the ESDM in all natural caretaking routines & play periods with their child. Parents are taught & coached on 1 aspect of the ESDM each week in the clinic session, & then practice it at home daily in natural family routines & play.
  Phase 2: each child in the ESDM will receive 25 hrs. a week of ESDM intervention in their homes, 50 wks. a year, for 2 years. 20 hrs. weekly will be delivered by trained interventionists (ITs); 5 hrs. weekly will be delivered by parents. (ITs) will provide ten 2 hour teaching episodes involving play activities per week in the home. Parents will continue to deliver the ESDM in natural family routines & play activities. In addition, each child will receive additional services through public services, or other therapies that the parents may choose, for several more hrs. per week.
  Interventions: Behavioral: Early Start Denver Model
- 2 Standard Care available in the Community (Other): Any intervention that were available and that families accessed in their communities
  Interventions: Behavioral: Standard community care

INTERVENTIONS:
Behavioral: Early Start Denver Model — Phase 1 of ESDM intervention: 12 weekly, 1 to 1.5 hr. sessions focused on teaching & coaching parents to use the ESDM in all natural caretaking routines & play periods with their child. Parents are taught & coached on 1 aspect of the ESDM each week in the clinic session, & then practice it at home daily in natural family routines & play.
  Phase 2: each child in the ESDM will receive 25 hrs. a week of ESDM intervention in their homes, 50 wks. a year, for 2 years. 20 hrs. weekly will be delivered by trained interventionists (ITs); 5 hrs. weekly will be delivered by parents. (ITs) will provide ten 2 hour teaching episodes involving play activities per week in the home. Parents will continue to deliver the ESDM in natural family routines & play activities. In addition, each child will receive additional services through public services, or other therapies that the parents may choose, for several more hrs. per week.
  Other Names: intensive intervention for infants and toddlers with autism and ASD; autism treatment; PDD NOS; University of California, Davis; Sally Rogers; University of Washington and early autism intervention; University of Michigan and early intervention
  Arms: 1 Early Start Denver Model
Behavioral: Standard community care — Treatment and interventions, chosen by families, meeting current standards of community intervention for toddlers with autism and ASD
  Other Names: Current, standard community based intervention for toddlers with autism; intensive intervention for infants and toddlers with autism and ASD; autism treatment; PDD NOS; University of California, Davis; Sally Rogers; University of Washington and early autism intervention; University of Michigan and early intervention
  Arms: 2 Standard Care available in the Community

SUMMARY:
Goals of the current project: (1) Does the Early Start Denver Model experimental intervention for toddlers with autism reduce disability associated with autism significantly more than standard community interventions?; and (2) What environmental, child, and biological characteristics mediate and moderate intervention response and outcomes at age 4?

DETAILED DESCRIPTION:
Thanks to the development of better diagnostic tools and a greater level of professional education, autism is being identified in two year olds and in even younger children, with such early diagnosis justified by the rationale that the earlier intervention begins, the better the outcomes may be. However, there are no published outcome data on intervention models or effectiveness for children who begin intervention by or before 24 months. Furthermore, some teaching procedures considered appropriate for older children, (e.g., 40 hours per week of adult-directed intervention, much repetitive practice while sitting at a table (Lovaas, 2002), 1987) are considered developmentally inappropriate for toddlers (Sandall, McLean, & Smith, 2000).

Dawson and Rogers have implemented a feasibility study of a intervention designed for toddlers with autism using a randomized controlled design. The approach involves a relationship-based frame to accomplish developmentally based objectives using naturalistic application of applied behavior analytic principles. The approach fuses the Denver Model (Rogers, Hall, Osaki, Reaven, & Herbison, 2000) and Pivotal Response Training (Koegel, Koegel, & Carter, 1999), and is delivered 1:1 for 25 or more hours per week to 24 toddlers with autism for a two year period. The contrast group receives standard community based intervention. Preliminary results demonstrate large and significant group effects after only 12 months and considerable variability of intervention outcomes in both groups.

All families will be referred to the appropriate community service programs, if they have not been referred previously.

ELIGIBILITY:
Inclusion criteria: (1) 12-24 months of age at the time of telephone screening and living within 60 minutes of the university clinic; (2) ambulatory; (3) unimpaired hand use; (4) parent agreement to have a caregiver present during all home sessions; (5) attendance at all intake sessions; (6) permission to videotape evaluations and ESDM treatment; (7) English as one primary language of the parent; (8) unimpaired hearing and vision; (9) developmental quotient of 35 or higher on the Mullen Scales of Early Learning (MSEL); and (10) meets all of these ASD diagnostic criteria: (a) Autism Diagnostic Observation Scale for Toddlers (ADOS-T) cutoff score of 12 if child produces no words or 10 if child produces some words; (b) agreement by two experienced psychologists that ASD is present; and that child meets DSM-IV criteria for Autistic Disorder or Pervasive Developmental Disorder Not Otherwise Specified (PDDNOS). 5,7,8 Exclusion criteria: (1) serious parental substance abuse; (2) parental self-report of bipolar disorder or psychosis; (3) known genetic syndromes; (4) serious medical conditions (e.g., encephalitis, concussion, seizure disorder); (5) significant sensory impairment; (6) birth weight <1600 grams and/or gestational age < 34 weeks; (7) history of intraventricular hemorrhage; (8) known exposure to neurotoxins (including alcohol, drugs); (9) non-English-speaking parents; and for the ESDM-assigned group only, (10) current enrollment in an intensive, 1:1 delivered behavioral intervention of more than 10 hours per week. There was no other restrictions on additional community-based treatment.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sally J Rogers, Ph.D., Principal Investigator — UC Davis MIND Institute
Locations (1):
- UC Davis Mind Institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data from primary analyses are available on NDA.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: September 2019 - September 2021
Access Criteria: access data via NDA: https://nda.nih.gov request other materials from PI srogers@ucdavis.edu

REFERENCES:
- [Derived] Rogers SJ, Estes A, Lord C, Munson J, Rocha M, Winter J, Greenson J, Colombi C, Dawson G, Vismara LA, Sugar CA, Hellemann G, Whelan F, Talbott M. A Multisite Randomized Controlled Two-Phase Trial of the Early Start Denver Model Compared to Treatment as Usual. J Am Acad Child Adolesc Psychiatry. 2019 Sep;58(9):853-865. doi: 10.1016/j.jaac.2019.01.004. Epub 2019 Jan 24. PMID 30768394
- [Derived] Zhou V, Munson JA, Greenson J, Hou Y, Rogers S, Estes AM. An exploratory longitudinal study of social and language outcomes in children with autism in bilingual home environments. Autism. 2019 Feb;23(2):394-404. doi: 10.1177/1362361317743251. Epub 2017 Dec 13. PMID 29237275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were recruited from pediatricians, developmental disability settings, and university website postings using IRB-approved materials.
Groups:
- 1 Early Start Denver Model: Phase 1 of ESDM intervention: 12 weekly, 1 to 1.5 hr. sessions focused on teaching & coaching parents to use the ESDM in all natural caretaking routines & play periods with their child. Parents are taught & coached on 1 aspect of the ESDM each week in the clinic session, & then practice it at home daily in natural family routines & play.
  Phase 2: each child in the ESDM was assigned to receive 20 hrs. a week of ESDM intervention in their homes, 50 wks. a year, for 2 years by trained interventionists (ITs). Parents delivered ESDM in natural family routines & play activities as they chose. In addition, children received additional public and or private services as their families chose.
  Both phases followed published treatment manuals and all treatment was supervised by professionals with ESDM certification.
Period: Overall Study
Arm/Group | 1 Early Start Denver Model | 2 Standard Care Available in the Community
Started | 55 (1 enrollment) | 63 (1 enrollment)
Completed | 45 (45 - final participant assessment completed) | 36 (36 - final assessment completed)
Not Completed | 10 | 27
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 7 | 27

BASELINE CHARACTERISTICS:
Groups:
- Standard Care Available in the Community: Standard community care: Treatment and interventions, chosen by families, meeting current standards of community intervention for toddlers with autism and ASD
- Total: Total of all reporting groups
Arm/Group | Early Start Denver Model | Standard Care Available in the Community | Total
Number analyzed (Participants) | 55 | 63 | 118
Age, Continuous [Mean (Standard Deviation); unit: months] | 20.58 (3.37) | 20.70 (3.21) | 20.64 (3.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 41 | 51 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 10 | 16
  Not Hispanic or Latino | 45 | 49 | 94
  Unknown or Not Reported | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 37 | 43 | 80
  More than one race | 8 | 9 | 17
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 55 | 63 | 118

OUTCOME MEASURES:

1. Primary Outcome: Language Age Equivalent
Description: Composite language measure consisting of an average of the Expressive Language and the Receptive Language age equivalent scores from the Mullen Scales of Early Learning.The Mullen Scales of Early Learning (MSEL) is a developmental test with five subscales: gross motor, visual reception, fine motor, receptive language, and expressive language. The lower the score on this scale, the more immature the ability; the higher the score, the more mature the ability. Measurements were taken at baseline, 6 months, 12 months, and 24 months and a hierarchical longitudinal growth curve approach used to calculate overall rate of growth during the 24 month period.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: language age in months
Arm/Group | 1 Early Start Denver Model | Standard Care Available in the Community
Number analyzed (Participants) | 55 | 63
language age in months | 39.59 (15.31) | 36.09 (14.52)
Statistical Analysis 1: Comparison: 1 Early Start Denver Model vs Standard Care Available in the Community; We used a generalized linear mixed model (GLMM). Change-over-Time was modeled as a linear within-subject effect of time across all observed data for each participant. We fit splines to manage the differing lengths of time in parent-training versus direct treatment. In all analyses, site was included as a categorical covariate to account for potential differences. Effect sizes were reported following Cohen's recommendations as f2; Test type: Other — Non- equivalence; p = .03, Mixed Models Analysis; slope difference = 1.01

2. Secondary Outcome: Overall Developmental Quotient (DQ)
Description: Overall DQ was calculated by averaging the Time 1 (baseline) age equivalence scores of the two language and two nonverbal subtests from the Mullen Scales of Early Learning (MSEL), dividing by child age in months, and multiplying by 100 to create a quotient score, in order to capture the full range of variability of the sample, since many children fell below the basal standard score. The Mullen Scales of Early Learning (MSEL) is a developmental test with five subscales: gross motor, visual reception, fine motor, receptive language, and expressive language. Gross motor score was not used for the calculations. The lower the score on this scale, the more immature the ability; the higher the score, the more mature the ability. Measurements were taken at baseline, 6 months, 12 months, and 24 months and a hierarchical longitudinal growth curve approach used to calculate overall rate of growth during the 24 month period.
Time Frame: 24 months
Measure: Mean (Standard Error); unit: developmental quotient
Arm/Group | 1 Early Start Denver Model | Standard Care Available in the Community
Number analyzed (Participants) | 55 | 63
developmental quotient | 83.09 (26.12) | 79.14 (25.58)

3. Secondary Outcome: Adaptive Behavior Age Equivalent Scores
Description: Adaptive behavior age equivalent was characterized by averaging the means of the age equivalents in months of the four domain scores from the Vineland Adaptive Behavior Scales - Second edition (VABS) because the manual does not provide developmental ages corresponding to total scores that could be used to construct quotient scores. Data were provided by parents who were not naïve to group assignment. The Vineland Adaptive Behavior Scales 2 provide a standardized measure of adaptive behavior in four domains: motor, language, social, and activities of daily living. Information is gathered from parents via parent questionnaire. The lower the score on each domain score and the overall score, the more immature the ability; the higher the score, the more mature the ability. Measurements were taken at baseline, 6 months, 12 months, and 24 months and a hierarchical longitudinal growth curve approach used to calculate overall rate of growth during the 24 month period.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: months
Arm/Group | 1 Early Start Denver Model | Standard Care Available in the Community
Number analyzed (Participants) | 55 | 63
months | 39.76 (12.07) | 36.69 (14.32)

4. Secondary Outcome: Autism Severity
Description: Autism severity was calculated using the Calibrated Severity Scores, derived by using tables in publications by Gotham, Pickles, & Lord( 2012) (Esler, Bal, Guthrie, Weismer, and Lord, 2015). We identified the severity score listed in the CSS table that was associated with a subject's ADOS-2 total score for the ADOS module that was administered to each subject at each of four time points - at entry into the project, and 6 months, 12 months, and 24 months after enrollment. The ADOS Calibrated Severity Score scale range is 1-10, with lower scores representing milder and less numerous symptoms and higher scores representing more severe and more numerous systems. Scores 1-3 represent few to no ASD symptoms, scores of 4-5 represent mild to moderate symptoms and concerns related to ASD, and scores of 6-10 represent moderate to severe symptom severity.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 2Standard Care Available in the Community: Standard Care available in the Community
  Standard community care: Treatment and interventions, chosen by families, meeting current standards of community intervention for toddlers with autism and ASD
Arm/Group | 1 Early Start Denver Model | 2Standard Care Available in the Community
Number analyzed (Participants) | 55 | 63
units on a scale | 6.69 (1.96) | 6.19 (2.52)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | 1 Early Start Denver Model | Standard Care Available in the Community
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/63
Other Adverse Events (participants affected / at risk) | 0/55 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT00698997/Prot_000.pdf